CLINICAL TRIAL: NCT05529563
Title: The Effect of Laparoscopic Sleeve Gastrectomy on Insulin Secretion Pattern in Morbidly Obese Patients With Acanthosis Nigricans
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shen Qu (Other)
Responsible Party: Sponsor-Investigator, Shen Qu, Principle investigator, Shanghai 10th People's Hospital
Organization: Shanghai 10th People's Hospital (Other)
Other Study IDs: Acanthosis Nigricans
Record Dates: First submitted 2022-09-02; First posted 2022-09-07 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Morbid Obesity; Acanthosis Nigricans; Insulin Resistance; Insulin Sensitivity; Bariatric Surgery Candidate
Keywords: Acanthosis nigricans; Morbid obesity; Insulin secretion pattern; Prolactin; Sleeve gastrectomy
MeSH Terms: conditions — Obesity, Morbid; Acanthosis Nigricans; Insulin Resistance

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- obesity without AN (OB group) and obesity with AN (AN group): LSG
  Interventions: Procedure: LSG

INTERVENTIONS:
Procedure: LSG — LSG

SUMMARY:
Acanthosis nigricans (AN) is increasing in its prevalence and is the most prevalent cutaneous manifestation in individuals with obesity. Insulin resistance or hyperinsulinemia is the main pathophysiological mechanism of obesity-related AN. However, the effect of laparoscopic sleeve gastrectomy (LSG) on insulin secretion pattern in Chinese morbidly obese patients with AN is unknown. In these study, the investigators aimed to explore the insulin secretion patterns in Chinese morbidly obese patients with Acanthosis nigricans (AN) and their alterations after LSG.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 to 65 years
* BMI equal or greater than 35 kg/m2
* completed a 75-g OGTT and insulin release assay
* eligible for the 12-month follow-up.

Exclusion Criteria:

* severe liver and renal dysfunction, preexisting heart disease, malignancy, or endocrine diseases such as pituitary adenoma and hypogonadism
* mental illness
* genetic disease
* current or previous treatment that might affect the sex hormones and insulin secretion
* gestation or lactation
* loss to follow-up, or withdrawal from the study
* unable to understand and comply with the study protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who met the inclusion and exclusion criteria were enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 138 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
Obesity | 2017-2023
  It was defined as BMI ≥ 28 kg/m2 according to the diagnostic criteria for obesity in a Chinese population.
A quantitative scale of Acanthosis Nigricans (AN) | 2017-2023
  0-absent: not detectable on close inspection; 1-present: clearly present on close visual inspection, not visible to the casual observer, extent not measurable; 2-mild: limited to the base of the skull, does not extend to the lateral margins of the neck (usually <3 inches in breadth); 3-moderate: extending to the lateral margins of the neck (posterior border of the sternocleidomastoid, usually 3-6 inches), should not be visible when the participant is viewed from the front; 4-severe: extending anteriorly (>6 inches), visible when the participant is viewed from the front.
Insulin secretion patterns | 2017-2023
  they were derived from the peak time of insulin secretion during OGTT: Type I (peak time at 30 or 60 min) and Type II (peak time at 120 or 180 min).

SECONDARY OUTCOMES:
BMI | 2017-2023
  It was calculated as weight (kg) divided by squared height (meters).
a 2-h 75-g oral glucose tolerance test (OGTT) | 2017-2023
  It was performed after an overnight fasting in each patient pre- and 12 months pro-LSG, and blood samples were taken at 0, 30, 60, 120, and 180 min to determine the concentrations of plasma glucose and insulin.
HOMA-IR | 2017-2023
  It was calculated as FPG (mmol/L)×FINS (mU/L)/22.5 (24).
Insulin sensitivity | 2017-2023
  It derived from the OGTT was estimated by the oral glucose insulin sensitivity (OGIS) index
Insulinogenic index (IGI) | 2017-2023
  It was calculated as :(insulin30min-insulin0min)/ (glucose30min-glucose0min).
the disposition index (DI) | 2017-2023
  It was calculated as IGI/HOMA-IR.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Tenth People's Hospital, Shanghai, China